CLINICAL TRIAL: NCT00825513
Title: Monocular Study to Evaluate the Safety and Effectiveness of the Akreos™ Toric IOL When Used to Correct Primary Aphakia With the Reduction of Astigmatism
Brief Title: Safety and Effectiveness of the Akreos Toric Intraocular Lens.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 566
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Cataract; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Akreos Toric (Experimental): Akreos Toric Intraocular Lens
  Interventions: Device: Akreos Toric IOL
- Akreos Advanced (Active Comparator): Akreos Advanced Optics Aspheric Intraocular Lens (Akreos AO)
  Interventions: Device: Akreos Advanced Optics Aspheric Intraocular Lens (Akreos AO)

INTERVENTIONS:
Device: Akreos Toric IOL — Lens implant following cataract surgery
  Arms: Akreos Toric
Device: Akreos Advanced Optics Aspheric Intraocular Lens (Akreos AO) — Lens implant following cataract surgery
  Arms: Akreos Advanced

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Akreos Toric IOL following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to provide written consent on the EC approved Informed Consent form.
* Subjects must require a lens power from 15 to 30 diopters.

Exclusion Criteria:

* Subjects with any anterior segment pathology for which extracapsular phacoemulsification cataract surgery would be contraindicated.
* Subjects with corneal pathology potentially affecting topography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-02; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Reduction of cylinder, Lens axis misalignment as determined by a photographic method. | 32 months

SECONDARY OUTCOMES:
Lens misalignment as determined by postoperative manifest refraction and vector analysis. | 32 months

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Brenger, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Dept. of Clinical Sciences/ Ophthalmology Umea University Hospital, Umeå, Sweden